CLINICAL TRIAL: NCT03946891
Title: Nebulized Furosemide in Premature Infants With Bronchopulmonary Dysplasia - A Cross Over Pilot Study of Its Efficacy and Safety
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The study was stopped due to lack of study staff and inability to enroll subjects into the study due to restrictive inclusion criteria.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-01665
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Premature Birth; Premature Infant
MeSH Terms: conditions — Premature Birth | interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: Inhaled Furosemide
- Arm B (Experimental)
  Interventions: Drug: Intravenous Furosemide

INTERVENTIONS:
Drug: Inhaled Furosemide — Subjects in the A arm will receive 1 mg/kg of inhaled furosemide Q 24 hours for 3 days. This will be followed by a washout period of a day followed by 1 mg/kg of intravenous furosemide Q 24 hours for 3 days.
  Other Names: furosemide
  Arms: Arm A
Drug: Intravenous Furosemide — Subjects in the B arm will receive 1 mg/kg of intravenous furosemide Q 24 hours for 3 days followed by a washout period, which is then followed by 1 mg/kg of inhaled furosemide Q 24 hours for 3 days.
  Arms: Arm B

SUMMARY:
This is a prospective,randomized, cross over study comparing the efficacy and safety of nebulizedfurosemide with Intra Venous (IV)furosemide in preterm infants who areventilator-and oxygen dependent. Reviewing the patient census on Neo data by the Sub Investigator will identify the potential subjects. Subject will be randomized to either A arm or B arm. Subjects in the A arm will receive 1 mg/kg of inhaled furosemideQ 24 hours for 3 days. This will be followed by a washout period of a day followed by 1mg/kg of intravenous furosemide Q 24 hours for 3 days. Subjects in the B arm will receive 1 mg/kg of intravenous furosemide Q 24 hours for 3 days followed by a washout period, which is then followed by 1 mg/kg of inhaled furosemide Q 24 hours for 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are born prematurely at<34 weeks of gestation
* Subjects who are at least 14days old, on Oxygen and mechanical ventilation.
* Radiologic evidence of pulmonary parenchymal disease
* The NICU medical team to start furosemide administration as a part of the routine clinical management

Exclusion Criteria:

* Subjects who have received any diuretics;IV or PO for 48 hoursbefore the study initiation
* Subjects with congenital heart disease withR-L shunts.
* Subjects with acute sepsis.
* Subjects with kidney diseasedefined by creatinine > 1mg/dl or oliguria, defined as urine output < 0.6 ml/kg/hour
* Subjects with necrotizing enterocolitis (NEC)or suspected NEC
* Subjects with congenital malformations.Subjects who are receiving steroids, or have received steroids in the last 7 days(patients need to be off steroids for at least 7 days).

Ages: 0 Years to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Daily percent change from pre-treatment FiO2 requirement measurement. | days 1, 2, 3, 5, 6, and 7
  Measurements will be taken twice within a two-hour window before and after treatment as applicable. On baseline day and the washout day, two measurements will be also taken within the two-hour window to compute percent change for the day

CONTACTS AND LOCATIONS:
Overall Officials: Melodi Pirzada, MD, Principal Investigator — New York Langone Medical Center
Locations (1):
- New York University School of Medicine, New York, New York, United States